CLINICAL TRIAL: NCT03806712
Title: Comprehensive Study of Social Representation of Platelet Transfusion in Patients Followed for Advanced Hematological Malignancies (R-PLQ)
Acronym: R-PLQ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/413
Record Dates: First submitted 2018-12-30; First posted 2019-01-16 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Platelet Transfusion; Hematological Malignancy; Palliative Care
Keywords: social representation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patient: patient with advanced, non curative hematological malignancies multi method questionary, at least 1 hour per patient
  Interventions: Other: multi method questionary (developped by De Rosa, in 1995 and 2014)
- hematologist: medical practitioner of platelet transfusion multi method questionary, at least 1 hour per hematologist
  Interventions: Other: multi method questionary (developped by De Rosa, in 1995 and 2014)
- Nurses: nurses working in hematology, practicing platelet transfusion multi method questionary, at least 1 hour per nurse
  Interventions: Other: multi method questionary (developped by De Rosa, in 1995 and 2014)

INTERVENTIONS:
Other: multi method questionary (developped by De Rosa, in 1995 and 2014) — questions from an association network according to the subject and the grounded theorise (Glasser and Strauss)

SUMMARY:
Limited data is available for end of life care in hematologic malignancies, moreover with thrombocytopenic patients. Thrombopenia is a frequent complication, specific of bone marrow involvement in those diseases or its treatments. Yet, a few studies was interested in, whereas platelet transfusion is the only treatment indicated. As it represent a scarce, limited resource, the ethical principles are in conflict in this setting and there's a lack of recommendation. The final decision is take by the clinician and his patient, but no study exist in representation of the two parts. We provide a qualitative study to understand what this decision is made of.

ELIGIBILITY:
Inclusion Criteria:

* major patient
* patient with advanced hematological malignancies
* patient transfused in platelet regularly (3 time at least in last month)
* medical practioner, hematologist, prescribing platelet transfusion at least one per week.
* nurse working in hematology, practicing platelet transfusion at lest one peer week.

Exclusion Criteria:

* minor patient
* non communicant patient
* non transfused platelet patient
* non voluntary patient or hematologist or nurses
* non graduated hematologist

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with advanced hematological malignancies, transfused in platelet regulary, hematologist's nurses who practice platelet transfusion and hematologist who prescribe the transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
measure the impact of social representation on platelet transfusion practice | 3 months
  inner core and peripheral items of platelet transfusion of each participant will be collected until reaching saturation, it's to say that the repetition of some terms will be measured between each interview thank's to a questionnaire of at least two principals opened questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Moracchini, Besançon, France

IPD SHARING:
Plan to Share IPD: No
interview will be registered then transcribe on professional computer ans accessible only by the investigator and collaborators.

REFERENCES:
- [Background] McGrath P, Leahy M. Catastrophic bleeds during end-of-life care in haematology: controversies from Australian research. Support Care Cancer. 2009 May;17(5):527-37. doi: 10.1007/s00520-008-0506-1. Epub 2008 Sep 23. PMID 18810505
- [Background] McGrath P, Holewa H. Special considerations for haematology patients in relation to end-of-life care: Australian findings. Eur J Cancer Care (Engl). 2007 Mar;16(2):164-71. doi: 10.1111/j.1365-2354.2006.00745.x. PMID 17371426
- [Background] Jeoffrion C, Dupont P, Tripodi D, Roland-Levy C. [Social representations of illness: Comparison of "expert" knowledge and "naive" knowledge]. Encephale. 2016 Jun;42(3):226-33. doi: 10.1016/j.encep.2015.12.007. Epub 2016 Jan 12. French. PMID 26796561